CLINICAL TRIAL: NCT07006844
Title: Comparison of Analgesic Efficacy of Fascia Transversalis Plan Block and Caudal Epidural Block in Pediatric Patients Undergoing Orchiopexy. Our Study, it Was Planned to Compare the Postoperative Analgesic Efficacy of Routinely Applied Fascia Transversalis Plan Block and Caudal Epidural Block for Analgesia After General Anesthesia in Pediatric Patients Undergoing Orchiopexy (Unilateral) According to the Surgery and Suitability of the Patient and the Competence of the Anesthesiologist
Brief Title: Comparison of Analgesic Efficacy of Fascia Transversalis Plan Block and Caudal Epidural Block in Pediatric Patients Undergoing Orchiopexy
Status: Not yet recruiting | Type: Observational
Sponsor: Prof. Dr. Cemil Tascıoglu Education and Research Hospital Organization (Other)
Responsible Party: Principal Investigator, Ece Ozcan, research assistant, Prof. Dr. Cemil Tascıoglu Education and Research Hospital Organization
Other Study IDs: E-48670771-514.99-273708811...
Record Dates: First submitted 2025-05-28; First posted 2025-06-05 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-05

CONDITIONS: Orchiopexy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- fascia transversalis plan block group: In fascia transversalis plan block, it is aimed to block the ilioinguinal and iliohypogastric nerves by injecting local anesthetic into the fascia transversalis plane under ultrasound guidance. It is a preferred method for analgesia of inguinal and lower abdominal surgeries
- Caudal epidural block group: Caudal epidural block is a regional anesthesia technique performed by administering local anesthetic or analgesic drugs into the epidural space through the sacral hiatus. It is frequently used in urogenital, rectal, inguinal and lower extremity surgeries.

SUMMARY:
Orchiopexy is a surgery with a high frequency in the pediatric population. The use of regional anesthesia techniques has become widespread and its importance has increased in order to provide more effective and prolonged perioperative analgesia, as well as to prevent the side effects of opioids such as respiratory depression and to reduce systemic analgesic consumption. In this study, it was planned to compare the postoperative analgesic efficacy of routinely applied fascia transversalis plan block and caudal epidural block for analgesia after general anesthesia in pediatric patients undergoing orchiopexy (unilateral) according to the surgery and suitability of the patient and the competence of the anesthesiologist.

ASA I-II, patients who will undergo unilateral orchiopexy under general anesthesia, patients between the ages of 1-7 years, who have no contraindications for block application, and whose participation in the study is accepted by their legal guardian will be included in the study. After induction of general anesthesia and ensuring airway safety with a laryngeal mask, one of the regional anesthesia methods (fascia transversalis plan block or caudal epidural block) deemed appropriate for the patient is applied by the specialist of the room before the surgical incision. Postoperative analgesic needs of the patients and FLACC score will be evaluated at 30 minutes, 1, 2, 4, 6, 12 and 24 hours postoperatively.

ELIGIBILITY:
Inclusion Criteria:

ASA I-II, patients who will undergo unilateral orchiopexy under general anesthesia patients between the ages of 1-7 years, who have no contraindications for block application, and whose participation in the study is accepted by their legal guardian will be included in the study.

Exclusion Criteria:

Lack of consent by the patient's legal guardian, contraindications for block (bleeding diathesis, regional infection, neuromuscular disease), patients over 7 years of age

Ages: 1 Year to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: ASA I-II, patients who will undergo unilateral orchiopexy under general anesthesia, patients between the ages of 1-7 years
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-06-07 (Estimated); Primary Completion 2025-12-21 (Estimated); Study Completion 2026-01-07 (Estimated)

PRIMARY OUTCOMES:
FLACC (The Faces, Legs, Activity, Cry and Consolability) pain scoring | Postoperative 30 minutes 1, 2, 4, 6, 12 and 24 hours
  The Face, Legs, Activity, Crying, and Consolability (FLACC) scale is an observational pain scale. It is widely used in the pediatric population to assess pain in infants and children who cannot verbally express their pain. [1] Instead, the FLACC scale was developed to help patients understand their pain experience by observing facial expressions and behavioral patterns to enable the provision of effective pain intervention.

SECONDARY OUTCOMES:
Postoperative analgesic needs | Postoperative 30 minutes 1, 2, 4, 6, 12 and 24 hours
  Postoperative 30 minutes 1, 2, 4, 6, 12 and 24 hours analgesic consumption will be recorded

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Okur O, Tekgul ZT, Erkan N. Comparison of efficacy of transversus abdominis plane block and iliohypogastric/ilioinguinal nerve block for postoperative pain management in patients undergoing inguinal herniorrhaphy with spinal anesthesia: a prospective randomized controlled open-label study. J Anesth. 2017 Oct;31(5):678-685. doi: 10.1007/s00540-017-2378-3. Epub 2017 Jun 14. PMID 28616651
- [Result] Oksuz G, Arslan M, Urfalioglu A, Guler AG, Teksen S, Bilal B, Oksuz H. Comparison of quadratus lumborum block and caudal block for postoperative analgesia in pediatric patients undergoing inguinal hernia repair and orchiopexy surgeries: a randomized controlled trial. Reg Anesth Pain Med. 2020 Mar;45(3):187-191. doi: 10.1136/rapm-2019-101027. Epub 2020 Jan 5. PMID 31907294